CLINICAL TRIAL: NCT00048529
Title: Study of T900607-Sodium in Subjects With Previously Treated Gastric Cancer or Adenocarcinoma of the Esophagus
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Tularik (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-607-006
Record Dates: First submitted 2002-11-01; First posted 2002-11-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Gastric Cancer; Esophageal Neoplasms
Keywords: adenocarcinoma of the esophagus
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Adenocarcinoma Of Esophagus

INTERVENTIONS:
Drug: T900607-sodium intravenous

SUMMARY:
This is a clinical research study of T900607-sodium to determine if it is effective and safe in treating gastric cancer and adenocarcinoma of the esophagus. Patients will be treated on a weekly basis with an intravenous injection of the study drug.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of gastric cancer or adenocarcinoma of the esophagus
* Subjects must have received 1-2 regimens of prior chemotherapy
* At least 18 years of age
* Bidimensionally measurable disease amenable to CT scanning. At least one lesion must be least 1 X 1 cm in size.
* Karnofsky performance status of at least 70%
* Estimated life expectancy of at least 12 weeks
* Females of childbearing potential must have a negative pregnancy test and agree to use an effective contraceptive
* Subject must be able to comply with study procedures and follow-up examinations.
* Signed written informed consent
* Lab Values (obtained ≤ 7 days prior to study enrollment):

  * ANC at least 1.5x10e9/L, * Platelet count at least 100x10e9/L,
  * Creatinine within 2 times upper limit of normal * AST and ALT within 5 times upper limit of normal
  * Bilirubin within 1.5 times upper limit of normal
  * Albumin great than 2.5 g/dL

Exclusion Criteria

* Severe, concurrent disease, infection or co-morbidity that, in the judgment of the investigator, would make the subject inappropriate for enrollment
* NYHA Class III/IV cardiac disease, left ventricular ejection fraction (LVEF) of <50%, or acute anginal symptoms
* Patients who have received any investigational agent within 4 weeks of enrollment
* Patients who are pregnant or breast-feeding
* History of prior malignancy other than gastric cancer or adenocarcinoma of the esophagus within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* History of central nervous system metastases or carcinomatous meningitis
* Major surgery within 4 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Boyd, Study Chair
Locations (5):
- United States (5):
  - Pacific Oncology Associates, Los Gatos, California
  - Scripps Health Center, San Diego, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Ireland Cancer Center, Cleveland, Ohio